CLINICAL TRIAL: NCT01466413
Title: A Phase 1B Study to Assess the Safety and Efficacy of Two Formulations of ELAPR Compared to Restylane® Vital Light Following Repeat Implants in the Upper Arm Dermis
Brief Title: Two Formulations of ELAPR Compared to Restylane® Vital Light Following Repeat Implants in the Upper Arm Dermis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elastagen Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: ELAPR P1B
Record Dates: First submitted 2011-09-18; First posted 2011-11-08 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Intrinsic Aging of Skin
Keywords: Intrinsic Aging of Skin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane (Experimental): Patients with an even subject identification number (SIN) (02, 04, 06, 08, 10, 12, 14, 16) will have ELAPR to the right arm and the control to the left, where patients with an odd subject identification number (01, 03, 05, 07, 09, 11, 13, 15) will have the ELAPR to the left arm and the control to the right.
  Patients will receive either device ELAPR002c or ELAPR002e. This will alternate to minimise bias between the right and left arms.
  The first group of eight patients (01 - 08) will have their biopsy performed at day 169. The second group of eight patients (09 - 16) will have their biopsy at day 85.
  Interventions: Device: Tropoelastin

INTERVENTIONS:
Device: Tropoelastin — Multiple intradermal implants comprising of three treatments, 3 weeks apart, each consisting of 16 injections in total, each 10mm apart in a grid formation over a 3cm x 3cm area of the mid to deep dermis of the medial aspect of the upper arm. Each injection will consist of 20-30ul of product delivered using a 30Gx¼" needle. Each subject will also receive Restylane® Vital Light (control) to the opposite arm following the same treatment regimen and using the same technique. The treatment will be administered on Day 1, 22 and 43.
  Other Names: Restylane Vital Light

SUMMARY:
This is an early phase study comparing two fixed dose of the study compound ELAPR and a Restylane® Vital Light (control), by multiple intradermal injections to a 3cm x 3cm area of the upper arm dermis. All subjects will receive three treatments, 3 weeks apart. Each treatment will consist of 16 injections in total, each 10mm apart in a grid formation over a 3cm x 3cm area of the mid - to deep dermis of the medial aspect of the upper arm. Each injection will consist of 20-30ul of product delivered using a 30Gx¼" needle.

DETAILED DESCRIPTION:
Each subject will also receive Restylane® Vital Light (control) to the opposite arm following the same treatment regimen and using the same technique. A 4mm skin biopsy will be taken from each of the implant sites from Cohort A subjects (including replacements) on Day 169, and from Cohort B subjects (including replacements) on Day 85. The biopsy will encompass the needle point tattoo at the centre of the implant site. The biopsy site will be closed with a single stitch followed by standard aftercare procedures with stitch removal 7 to 10 days later.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 50 years
* Male or Female
* Good general health status
* Able to give informed consent

Exclusion Criteria:

* Clinically significant abnormalities of haematology or biochemistry testing
* Bleeding diathesis
* anticoagulant drugs
* thrombocytopenia or clinically significant prolonged APTT or PT
* Chronic use of aspirin, other non-steroidal anti-inflammatory drugs or other anti-platelet agents
* History of keloid formation
* Systemic corticosteroids within last 12 weeks
* Diabetes or other metabolic disorders that may interfere with the subject's response to treatment in the opinion of the investigator
* Any serious medical condition which in the opinion of the investigator would have a strong possibility of requiring systemic corticosteroid medication
* Pregnancy/lactation
* Previously received Tropoelastin
* A history of anaphylaxis or allergic reactions including any known hypersensitivity to Hyaluronic acid or lidocaine
* Sensitivity to Restylane® Vital light or Restylane products
* Use of any other investigational product on the intended implant site in the previous 12 months.
* Sensitivity to topical local anaesthetic cream (EMLA®) or have the following conditions where EMLA is contraindicated: dermatitis, Methaemoglobinaemia, Glucose-6-phosphate dehydrogenase deficiency or "Mollusca Contagiosa"

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Assess the persistence and tissue compatibility with histopathology. | 26 weeks
  A 4mm skin biopsy will be taken from each of the implant sites from Cohort A subjects on Day 169, and from Cohort B subjects on Day 85.

SECONDARY OUTCOMES:
Assess the acute and chronic safety of ELAPR. | 26 weeks
  Biopsy at day 85 or day 169 depending on randomization

CONTACTS AND LOCATIONS:
Overall Officials: Carlos China, MBBS, Principal Investigator — Woolcock Institute Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Glebe, New South Wales, Australia